CLINICAL TRIAL: NCT02692807
Title: Arthroscopic Surgical Procedures Versus Sham Surgery for Patients With Femoroacetabular Impingement and/or Labral Tears. A Multicentre, International, Double-blinded Randomized, Controlled Trial.
Brief Title: Arthroscopic Surgical Procedures vs Sham Surgery for Patients With Femoroacetabular Impingement and/or Labral Tears.
Acronym: HIPARTI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: La Trobe University (Other); University of Aarhus (Other); Lund University (Other); University of Oxford (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, May Arna Risberg, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAR-1- 2016; 2015091 (Other Grant/Funding Number: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2024-05

CONDITIONS: Surgery
Keywords: hip arthroscopy; femoroacetabular impingement; exercise therapy after hip arthroscopy; rehabilitation after hip arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: The RCT part of the HIPARTI Study has 2 arms, but there is also a prospective longitudinal study of those who are either not willing to participate in the RCT, or where the study takes part in collaborating countries were there is ONLY the prospective longitudinal ongoing (Australia). This part of the study is the HARP study. The HIPARTI consists on one RCT trial with two parallel arms, and one prospective cohort, the HARP study.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is only for the RCT Study - the double-blinded study. The HARP study consists of only a prospective longitudinal study With same outcome measure and follow-ups; hence, given 3 arms. The below "Allocation" and "Number of Subjects" is ONLY for the RCT part of the study
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hip arthroscopy surgical procedures (HIPARTI Study) (Active Comparator): Surgery is performed under general anaesthesia. Traction and joint access is controlled by fluoroscopy. A diagnostic round in the central and peripheral compartment is performed. Labrum, cartilage, and other possible conditions are looked for and findings are documented. Any labral, chondral and bony pathology (cam or pincer) is treated. Labrum may be debrided, sutured, detached and refixed if needed to treat a pincer lesion. Labrum is secured with suture anchors. Pincer and cam resection is performed using an arthroscopic burr. Cartilage lesions maybe left untreated or treated with debridement or microfracture.
  Interventions: Procedure: Arthroscopic surgical procedures
- Sham surgery (HIPARTI Study) (Placebo Comparator): The same arthroscopic procedures as stated above are preformed, but no surgical interventions related to Cam, Pincer, or labral tear are performed, only diagnostic round in the central and peripheral compartment is performed. Labrum, cartilage, and other possible conditions are looked for and findings are documented.
  Interventions: Procedure: Arthroscopic surgical procedures
- Prospective Cohort (HARP Study) (Active Comparator): Those that are not willing to be included in the RCT (HIPARTI Study), will be asked if they are willing to be included in the prospective cohort, or ongoing in countries were ONLY the surgery is performed (Australia). They will sign an informed concent and will undergo surgical interventions as part of usual care. Outcomes collected and follow-ups will be the same as for the RCT (HIPARTI).
  Interventions: Procedure: Arthroscopic surgical procedures

INTERVENTIONS:
Procedure: Arthroscopic surgical procedures — See arm/group description of Arthroscopic surgery and sham surgery (HIPARTI). HARP: only arthroscopic surgery
  Other Names: Sham Surgery

SUMMARY:
The primary aim of this study is to determine the efficacy of hip arthroscopic surgery compared to a sham surgery (diagnostic arthroscopy only) for patients with symptomatic and radiological findings related to impingement (FAI) and/or labral tears using a randomized controlled design (HIPARTI Study: Primary aim and the main paper: primary end point: iHOT 1 year follow-up)).

Our main hypothesis is that surgical procedures of the hip will demonstrate greater efficacy than sham surgery (diagnostic hip arthroscopy only) for hip related quality of life (iHOT-33) after 1 year and at further (HIPARTI Study).

The secondary aim of this study is to establish modifiable risk factors associated with pain, function, work participation and quality of life over 1 year in people aged 18-50 years with hip impingement and/or labral tears diagnosed at hip arthroscopy. (HARP Study: A separate paper will be published with this main aim for the HARP Study) Long-term follow-ups for HIPARTI Study as well as HARP Study will be performed at 2, 5 and 10 years (secondary aims and separate papers).

DETAILED DESCRIPTION:
This is a multicenter, international, assessor and patient blinded clinical RCT with two groups (primary aim). the HIPARTI Study with The design of this trial conforms to the SPIRIT guidelines.

All patients with hip pain eligible for hip arthroscopy in our routine care pathways will be identified in our outpatient clinics. Consultant orthopedic surgeons will determine a patient's eligibility for the study (based on inclusion and exclusion criteria for the study) and members of their team introduce the study to the patients and refer them to the research coordinators for further information. Patients will be provided with oral and written information about the study and be introduced to our consent form. If interest continues the patient will be provided with further information and arrangements will be made for a baseline appointment for assessment and consenting.

The baseline assessment appointments will occur within one month of the initial approach. At the baseline appointment patients will meet with the research coordinator and the independent research assistant/tester (physical therapist) who will be the blinded tester. Patients will return their signed informed consent form and baseline questions completed. Those who are not willing to participate in the RCT (HIPARTI Study), will be asked if interested in being included in a prospective longitudinal cohort study including similar baseline and follow-up tests as those in the RCT (this will be the HARP Study with separate papers published). All patients in the HARP Study will undergo hip arthroscopy surgery. The Australian site will include most of their patients in the HARP Study, since the majority of orthopedic surgeons working privately will not participate in the HIPARTI Study. Data collection will be performed electronically for both the HIPARTI and the HARP Studies entering all data in the approved Checkware system (www.checkware.no).

Each collaborating center will apply to the ethical committee and the Data Inspectorate in each country/institution. Approval was confirmed for Oslo University Hospital (HIPARTI) and Australia (HARP Study) in January 2016.

Randomization (HIPARTI) will occur prior to surgery, after final eligibility is confirmed. Randomizations will be performed centrally using an automated computer generated system. Block randomization and stratification for each center will be performed.

All patients will undergo imaging (which may include CT scan or at least 1.5 Tesla magnetic resonance imaging MRI) prior to the surgical assessment as part of routine care. All patients will also undergo standardized radiographs of the hips and pelvis also as part of routine care. Plain radiographs will be examined for evidence of osteoarthritis as joint space narrowing, osteophytes, cysts and subchondral hypertrophy. Several radiographic measurements will be performed among them: the alpha angle and lateral center-edge angle will be determined for the presence of FAI. Radiographs will also be part of follow-ups.

Participating orthopedic surgeons will be asked to coordinate their waiting lists to ensure the hip arthroscopy patients are called for surgery in accordance with the study protocol. Ideally, patients will complete their baseline assessment as close to the randomized treatment as possible (within 1 months). In the event that surgery cannot be performed within 1 month after baseline assessment, the same questions and assessments completed at baseline will be completed again. The standard followed-ups at the 6 months and 1 year include primary and secondary outcomes. One year is the primary end point where randomization code will be broken according to a predefined published statistical protocol (HIPARTI).

At all follow-ups the research coordinator/independent tester will attend. At the 6 month follow-up an independent orthopedic surgeon will attend regularly and take care of patients who are not satisfied. The aim is to use the following criteria as subjective complaint: equal or worse than 10 points for the IHOT-33 score compared to baseline. All patients can withdraw without giving a reason at any time (stated in the consent form that all patients need to sign). An unblinded orthopedic surgeon will of course be able to have access to the medical record regarding performed procedures at any time if need for the health of the patient.

All patients (in both groups in the RCT (HIPARTI) as well as in the HARP study) will undergo a postoperative rehabilitation program based on the best available evidence. Each patient will be treated by physical therapists who will be trained and proficient in post-hip arthroscopy rehabilitation. Rehabilitation will be delivered a minimum of 8 sessions over 3-months and then once a month for the following three months. Details of rehabilitation are outlined in Appendix Rehabilitation. This contains a treatment algorithm to guide clinical reasoning and progression of treatment (manual therapy, exercises and education) through weeks 1-12.

Long term follow-ups will be performed at 2, 5 and 10 years Due to lack of studies published within this field: clinical relevant differences as well as changes within groups and SD are difficult to estimate. Our sample size calculations are based on primary outcome iHOT 33 at 1 year: estimated effect-size to 0.6 and a power of 90, will give 60 in each group, and with expected 15% dropout will give 138 patients in total. Electronic randomization lists will be generated, and estimations of inclusion rates per site are included. Statistical analysis procedures will be published and analysis performed prior to opening the group allocation when all patients are included and followed through to the 1 year follow-up (main outcome).

ELIGIBILITY:
Inclusion Criteria:

* hip pain during daily and/or spor t ing activities;
* intra-articular hip pain with radiological signs of FAI and/or labral tears eligible for hip arthroscopy (to be determined in a pragmatic fashion by the surgeon based on clinical examination and imaging
* the patient is able to give written informed consent and to participate fully in the interventions and follow-up procedures

Exclusion Criteria:

* pain that is not confirmed by physical examination of the hip
* evidence of preexisting osteoarthritis, defined as Tonnis grade >1, or less than 3mm superior joint space width on AP pelvic radiograph
* center edge angle on radiograph <25°; (v) previous known hip pathology such as Perthes' disease, slipped upper femoral epiphysis or avascular necrosis
* previous hip injury such as acetabular fracture, hip dislocation or femoral neck fracture
* previous hip surgery
* medical conditions complicating surgery (ASA 3); (ix) inflammatory joint disease (RA, Bechterew etc)
* physical inability to undertake testing procedures
* expected lack of compliance such as cognitive impairment, drug abuse or similar;
* inability to understand the written and spoken language of the treatment centre;
* contra-indications to placebo surgery, which will include large loose body, chondral flap >1cm2 detached at 3 sides, complete labral radial flap tear and labral bucket-handle tear with complete avulsion >1.5cm long

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool (IHOT-33) | Baseline, 6,12 an 24 months follow-ups - 1 year follow-up is main outcome
  Patient-reported outcome measure (PRO)

SECONDARY OUTCOMES:
Expectations of surgery | Baseline
  Questionnaire
HOOS - Hip Dysfunction and Osteoarthritis Outcome Score | Baseline, 6,12 an 24 months follow-ups - only in some study sites
  Patient-reported outcome measure (PRO) 5 subscales
ASES Arthritis Self-Efficacy Scale | Baseline, 6,12 an 24 months follow-ups
  Self-Efficacy Scale questionnaire
Tampa scale of Kinesiophobia | Baseline, 6,12 an 24 months follow-ups
  Fear of movement questionnaire
Hip Sports Activity Scale (HSAS) | Baseline, 6,12 an 24 months follow-ups
  Activity Level (type)
Work place Activity Limitation Survey (WALS) | Baseline, 6,12 an 24 months follow-ups
  Questionnaire (only for some of the study sites)- only in some study sites
Patient Specific Functional Scale | Baseline, 6,12 an 24 months follow-up
  Patient report on 3 specific activities and their limitations - only in some study sites
Measures of hip physical impairment: | Baseline, 6,12 an 24 months follow-ups
  Range of motion
Hip muscle strength | Baseline, 6,12 an 24 months follow-ups
  Dynamometer
Single leg squat performance | Baseline, 6,12 an 24 months follow-ups
  Performance tests - only in some study sites
Total Hip Replacement. | 1, 2, 5 and 10 years follow-up
  Data from the Norwegian National Joint Registry on total hip joint arthroplasty (or similar registries from the other countries)

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — Oslo University Hospital; Lars Nordsletten, MD, PhD, Study Director — Oslo University Hospital
Locations (2):
- LaTrobe University, School Allied Health, College of Science, Helath and Engineering, Melbourne, Victoria, Australia
- Division of Orthopedic Surgery, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data will be shared across the sites participating in the HIPARTI and the HARP Study, according to the protocol and the decisions made by the Advisory Committee